CLINICAL TRIAL: NCT03525990
Title: PRO-COM Project: Randomized-controlled Study Evaluating the Impact of Electronic Patient Reported Outcome (ePRO) Surveys on Patient-physician Communication and Quality of Life in Patients With Advanced Breast Cancer
Brief Title: Study Evaluating the Impact of Electronic Surveys on Patient-physician Communication and Quality of Life in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Vera Trommet (Other)
Responsible Party: Sponsor-Investigator, Dr. Vera Trommet, Principal Investigator, Klinikum Wels-Grieskirchen
Organization: Klinikum Wels-Grieskirchen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017/01
Record Dates: First submitted 2018-04-24; First posted 2018-05-16 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Breast Neoplasm Malignant Female
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Active Comparator): Quality of life questionnaires (electronic patient reported outcomes) to be filled out by the patients at every visit. Quality of life data is fully available for physicians. Paper-based questionnaire (EORTC QLQ-COMU26) at baseline, after three months and after six months.
  Interventions: Other: Questionnaires
- Control Arm (Placebo Comparator): Quality of life questionnaires (electronic patient reported outcomes) only to filled out by the patients at baseline, after three months and after six months. Quality of life data is hidden for physicians. Paper-based questionnaire (EORTC QLQ-COMU26) at baseline, after three months and after six months.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Quality of life questionnaires on iPads with CHES (Computer-based Health Evaluation System), paper-based questionnaire (EORTC QLQ-COMU26)

SUMMARY:
PRO-COM Project: Randomized-controlled study evaluating the impact of electronic patient reported outcome (ePRO) surveys on patient-physician communication and quality of life in patients with advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Stage IV breast cancer
* Start of a systemic anti cancer therapy: chemotherapy -/+ antibody therapy 1st until 3rd line (palliative), endocrine therapy or other therapy without limit
* Estimated life expectancy of minimum six months
* Signed informed consent
* No cognitive or speech impairments

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Patient-physician communication | Up to six months
  The communication between patient and physician will be assessed with EORTC QLQ-COMU26. Presumably some patients have privacy concerns with electronic questionnaires. The EORTC-COMU26 is the most important questionnaire in this study because it is needed for the primary endpoint. It contains sensitive questions about how the patient experiences the communication during the visit. In order to avoid patients not filling out the questionnaire due to privacy concerns or being afraid of giving an honest opinion and the physician could read it electronically, the EORTC QLQ-COMU26 is paper-based and the patients can hand them in in the study office.

SECONDARY OUTCOMES:
Quality of life assessment | Arm A: at every visit for six months; Arm B: at baseline, three months, six months
  Quality of life will be assessed electronically with EORTC QLQ-C30.
Frequency of discontinuations of therapy | Up to six months
  The frequency of discontinuations will be assessed based on medical reports.
Duration of communication between physician and patient | At baseline, three months, six months in both groups
  Physicians call the study office at the beginning and at the end of the consultation at baseline, three months and six months. They will record the duration of the consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Trommet, Dr., Principal Investigator — Klinikum Wels-Grieskirchen GmbH, 4. Interne
Locations (2):
- Austria (2):
  - A.ö. Krankenhaus St. Josef Braunau GmbH, Braunau am Inn, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Wels, Upper Austria

IPD SHARING:
Plan to Share IPD: No